CLINICAL TRIAL: NCT02083289
Title: A 28-day Double-masked, Randomized, Parallel-group, Active Controlled Study of ONO-9054 Ophthalmic Solution in Subjects With Ocular Hypertension (OHT) or Open-angle Glaucoma (OAG)
Brief Title: A 28 Day Study of ONO-9054 Ophthalmic Solution in Subjects With Ocular Hypertension (OHT) or Open-angle Glaucoma (OAG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-9054IOU003
Record Dates: First submitted 2014-03-06; First posted 2014-03-11 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Ocular Hypertension; Open Angle-glaucoma
Keywords: ONO-9054; ocular hypertension (OHT); Open angle-glaucoma (OAG); Glaucoma; Eye Diseases; Mild to moderate
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma; Eye Diseases | interventions — propan-2-yl 4-(6-(4-(2,5-difluorophenoxy)-3-hydroxybut-1-en-1-yl)-7-hydroxyoctahydro-2H-cyclopenta(b)oxepin-3-yl)butanoate; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm 1 (Experimental): ONO-9054 eye drop solution, 30 µg/mL (0.003%), once daily in both eyes, for 28 days.
  Interventions: Drug: ONO-9054
- Active Comparator Arm 2 (Active Comparator): Latanoprost eye drop solution, 0.005%, once daily in both eyes for 28 days.
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: ONO-9054
  Arms: Experimental Arm 1
Drug: Latanoprost
  Other Names: Xalatan®
  Arms: Active Comparator Arm 2

SUMMARY:
The primary objectives of this study are to compare the safety, tolerability, and mean change from baseline in diurnal intraocular pressure (IOP) of ONO-9054 30 µg/mL (0.003%) to latanoprost 0.005% following ocular instillation once every evening for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-85 (inclusive) with confirmed diagnosis of OHT or OAG
* Confirmed diagnosis of bilateral OHT or mild to moderate chronic OAG
* Able to undergo washout of all ocular drugs
* An IOP ≥ 24 mmHg at 8:00 AM and ≥ 21 mmHg at 10:00 AM in at least 1 eye; but < 36 mmHg in both eyes at both Day -5 and Day 1
* Central corneal thickness 500-620 µm at screening and Day -5 in both eyes
* Best corrected visual acuity (BCVA) of +0.7 Log Mar or better

Exclusion Criteria:

* Any history of severe ocular trauma in either eye at any time
* History of angle closure or ocular laser surgery within the past 3 months or any refractive surgery procedure within the past 6 months of Screening Visit in the study eye(s)
* Cataracts that prevent observation or photography of the fundus in either eye

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mean change in diurnal IOP (average of four time points) from baseline | 28 days
Evaluating the safety parameters per protocol | 28 days
  Physical and ocular examinations (tolerability, hyperemia, visual acuity, pupillometry, corneal thickness, aqueous cells and flare), vital signs, and safety laboratory evaluations

SECONDARY OUTCOMES:
Diurnal IOP | 28 days
Mean change from baseline in IOP at each measured time point | 28 days
Treatment response rates | 28 days
Percent change from baseline in IOP at each measured time point | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharmaceutical Co., Ltd., Study Director — Ono Pharmaceutical Co. Ltd
Locations (12):
- United States (12):
  - Los Angeles Clinical Site, Los Angeles, California
  - Mission Hills Clinical Site, Mission Hills, California
  - Newport Beach Clinical Site, Newport Beach, California
  - Pasadena Clinical Site, Pasadena, California
  - Petaluma Clinical Site, Petaluma, California
  - Morrow Clinical Site, Morrow, Georgia
  - Roswell Clinical Site, Roswell, Georgia
  - New York Clinical Site, New York, New York
  - High Point Clinical Site, High Point, North Carolina
  - Cranberry Township Clinical Site, Cranberry Township, Pennsylvania
  - Philadelphia Clinical Site, Philadelphia, Pennsylvania
  - Austin Clinical Site, Austin, Texas

REFERENCES:
- [Derived] Miller Ellis E, Berlin MS, Ward CL, Sharpe JA, Jamil A, Harris A. Ocular hypotensive effect of the novel EP3/FP agonist ONO-9054 versus Xalatan: results of a 28-day, double-masked, randomised study. Br J Ophthalmol. 2017 Jun;101(6):796-800. doi: 10.1136/bjophthalmol-2016-309023. Epub 2016 Sep 20. PMID 27649982